CLINICAL TRIAL: NCT07228429
Title: Quantification of Calcinosis Cutis Disease Burden in Patients With Systemic Sclerosis Using Computed Tomography Images
Brief Title: Quantification of Calcinosis Cutis Disease Burden Using Computed Tomography Images
Status: Not yet recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000040280; 1R01AR085316-01A1 (NIH)
Record Dates: First submitted 2025-11-12; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Systemic Sclerosis (SSc); Calcinosis Cutis
MeSH Terms: conditions — Scleroderma, Systemic; Calcinosis Cutis | interventions — sodium thiosulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Systemic sclerosis participants with calcinosis: SSc participants with calcinosis treated with sodium thiosulfate STS per SOC over 6 months.
  Interventions: Drug: Sodium Thiosulfate (STS)

INTERVENTIONS:
Drug: Sodium Thiosulfate (STS) — Calcinosis cutis treatment , Twice daily for 6 months

SUMMARY:
The main purpose of this study is to develop sensitive radiographic measurement techniques that can be used as outcome measures along with patient-reported outcome instruments in clinical trials of calcinosis cutis treatments, and potentially be used to assess disease course and treatment response in clinical practice. The goal is to test the performance of the software.

ELIGIBILITY:
Inclusion Criteria:

* Scleroderma/systemic sclerosis patient with diagnosed calcinosis cutis who will be clinically treated with STS as they would in clinical SOC care
* Must be ≥ 18 years old and meet the 2013 American College of Rheumatology criteria for the diagnosis of systemic sclerosis (diffuse or limited)
* Receiving clinical care at Yale clinics

Exclusion Criteria:

* Unable to provide informed consent
* Currently pregnant or nursing
* Patients with a calcinosis ROI >6cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with SSc with clinically apparent calcinosis cutis on physical exam will be recruited from Yale clinics.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Modified Mawdsley Calcinosis Questionnaire (mMCQ) | Baseline, 3 months and 6 months
  An 18-question survey with an overall score of 0-10; each individual question ranges from 0-10, scores are totaled and averaged to and divided by 18 to create the overall score. Higher scores indicate higher disability from calcinosis.
Calcinosis VAS | Baseline, 3 months and 6 months
  Used to measure the severity of calcinosis-related pain or symptoms. Scored 0-100 with higher scores indicate
CT imaging measure | Baseline, 3 months and 6 months
  BioImageSuite Web will be used to measure the CT scan volumes. The measurements are quantified using voxel annotation and built-in computation software. The volume of each scan will be recorded.

SECONDARY OUTCOMES:
Association between the change in the mMCQ scores and the CT imaging measures | Baseline, 3 months and 6 months
  Association between the change in the mMCQ scores and the CT imaging measures will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Monique Hinchcliff, MD, MS, Principal Investigator — Yale University
Locations (1):
- Yale Scleroderma Program, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No